CLINICAL TRIAL: NCT04133766
Title: Community-based Nutrition Program Effectiveness Evaluation in Afghanistan
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for the study withdrawn by sponsor after baseline data collected
Sponsor: FHI 360 (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Ministry of Public Health, Islamic Republic of Afghanistan (Unknown); UNICEF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1407870
Record Dates: First submitted 2019-10-18; First posted 2019-10-21 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Child Malnutrition; Breast Feeding; Nutrition
Keywords: Nutrition; Breastfeeding; Handwashing; Food security; Low and Middle Income Country; Infant and Young Child Feeding
MeSH Terms: conditions — Child Nutrition Disorders; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-Based Nutrition Package (Experimental): The Community-Based Nutrition Package (CBNP) is a multi-level intervention that comprises: advocacy and training for government stakeholders and employees; selection and training of master trainers who then cascade the training at provincial level; and selection and training of community-level Nutrition Mobilizing Teams. The Nutrition Mobilizing Teams then organize a 2-day community mobilization session in the catchment areas of each health post to develop a community nutrition plan, which is then implemented by community health workers and two additional volunteers under the mentorship of the Nutrition Mobilizing Teams and with the support of the community members that participated in the community mobilization session.
  Interventions: Behavioral: Community Based Nutrition Package (CNBP)
- Standard of care (No Intervention): Current standard of existing community health services.

INTERVENTIONS:
Behavioral: Community Based Nutrition Package (CNBP) — The Community-Based Nutrition Package (CBNP) is a multi-level intervention that comprises: advocacy and training for government stakeholders and employees; selection and training of master trainers who then cascade the training at provincial level; and selection and training of community-level Nutrition Mobilizing Teams. The Nutrition Mobilizing Teams then organize a 2-day community mobilization session in the catchment areas of each health post to develop a community nutrition plan, which is then implemented by community health workers and two additional volunteers under the mentorship of the Nutrition Mobilizing Teams and with the support of the community members that participated in the community mobilization session.
  Arms: Community-Based Nutrition Package

SUMMARY:
The study will be a mixed methods, two-arm, cluster-randomized controlled trial. The primary aim of this evaluation is to measure the effectiveness of the Community-Based Nutrition Package intervention on child feeding practices among parents/caregivers to children 6 to 23 months of age in Afghanistan.

DETAILED DESCRIPTION:
The study will be a mixed methods, two-arm cluster-randomized controlled trial (CRT). Health facilities eligible to implement the CBNP in their catchment areas will serve as the unit of implementation and be randomly allocated to treatment or control groups. For each health facility, up to four health posts, among the 6-10 health posts typically attached to a health facility, will be randomly selected. Households in communities served by selected health posts will be mapped and a list of households with eligible participants will generated from which a random sample will be selected. Structured questionnaires will be administered to separate samples of women with children 6-23 months of age at baseline then approximately 18 months later. Semi-structured, in-depth interviews will also be conducted with a sub-set of selected women and samples of their husbands and mothers-in-law at baseline and endline.

ELIGIBILITY:
Inclusion criteria:

* Married adult woman (all married women are considered adults in Afghanistan, regardless of age)
* Has a child between 6 and 23 months of age. For women with more than one living child between ages 6 and 23 months, questions will be asked regarding dietary experiences for the elder of the two. For twins or multiple order siblings, the eldest will be selected based on birth order.
* Resident in the household

Exclusion criteria:

No specific exclusion criteria.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4076 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Proportion of children ages 6-23 months who receive a minimum acceptable diet | 18 months
  Proportion of children ages 6-23 months who receive a World Health Organization-defined minimum acceptable diet

SECONDARY OUTCOMES:
Proportion of women who report initiating breastfeeding within one hour of delivery | 18 months
  Initiating breastfeeding within one hour of birth will be measured by asking the women/mother if she initiated breastfeeding within one hour after the baby was delivered
Proportion of women who report exclusive breastfeeding for the first six months of a baby's life | 18 months
  Exclusive breastfeeding is defined as giving infants only breastmilk, with no supplemental solid foods or liquids, including water. This measure is by self-reported practice from the mother and is constructed from questions about first liquids/feeds, all liquids taken prior to six months of age, and age of first solid food.
Food Insecurity Experience Score | 18 months
  The level of household food insecurity experience, and ordinal categorical measure with values ranging from 0 to 8, as measured using the United Nation's Food and Agriculture Organization's Food Insecurity Experience Survey (FIES).
Participation in household decision-making | 18 months
  The role of men and women in the household in terms of primary decision maker is examined by a set of 8 items adapted from the Demographic and Health Survey. Nominal categorical items record the primary decision-maker within the household for a number of important decisions, including health care seeking behavior, major and minor household purchases, and behaviors related to nutrition such as food acquisition, preparation and consumption.
Proportion of respondents who can name five critical times for washing hands to prevent disease transmission | 18 months
  Handwashing knowledge will be measured by asking respondents if they can name the five critical times for washing hands to prevent disease transmission. Those five times include: after using the toilet, before eating, before preparing food, before breastfeeding and after changing a baby's diaper/napkin (or cleaning the baby if a diaper/napkin isn't used).
Proportion of households with a handwashing facilities stocked with soap | 18 months
  Presence of a handwashing station/facility with soap within the home will be measured both through self-report and through direct observation by the data collector, if permission is given by the participant and/or head of household.

CONTACTS AND LOCATIONS:
Overall Officials: Said Iftekhar Sadaat, MD, MPH, Principal Investigator — Ministry of Public Health, Islamic Republic of Afghanistan
Locations (3):
- Afghanistan (3):
  - Not applicable - Community-Based, Ghazni
  - Not applicable - Community-Based, Herat
  - Not applicable - Community-based, Parwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 12 months of study completion
Access Criteria: Data will be made available without restriction.